CLINICAL TRIAL: NCT05520593
Title: Preoperative Oral Hydration in the Ambulatory Arthroplasty Population :A Single-Blinded Randomized Control Trial
Brief Title: Preoperative Oral Hydration in the Ambulatory Arthroplasty Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Jose Rodriguez, Professor of Clinical Orthopaedic Surgery, Hospital for Special Surgery, New York
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-2597
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Same-day Discharge; Length of Stay
Keywords: Carbohydrate Drink; Perioperative Fluids; Same-day Discharge; Total Joint Arthroplasty; Nausea; Vomiting; Same-day total hip arthroplasty; Same-day total knee arthroplasty
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complex Carbohydrate Drink Group (Experimental): The patients will drink a 400ml drink that contains 50g of complex carbohydrates, 3 hours prior to the surgery. The drink will be given once at the preoperative holding area. Patients are not allowed to eat solid foods after 12am the morning of surgery and can only drink clear fluids up to 3 hours prior to the surgery.
  Interventions: Dietary Supplement: Complex Carbohydrate Drink
- No-Complex Carbohydrate Drink Group (No Intervention): These patients will follow normal institutional preoperative fluid management guidelines, this consist of no solid foods after 12am the morning of surgery. Patients are allowed to drink clear liquids (water, clear fruit juices, coffee) from 12am the morning of surgery up to 3 hours prior to the surgery.

INTERVENTIONS:
Dietary Supplement: Complex Carbohydrate Drink — Patients will drink a complex carbohydrate drink 3 hours before surgery. Drink to be given at the preoperative holding area.
  Arms: Complex Carbohydrate Drink Group

SUMMARY:
The purpose of this study is to investigate if the consumption of a complex carbohydrate drink preoperatively, decreases the length of stay and causes for failure to launch in patients undergoing ambulatory total joint arthroplasty.

DETAILED DESCRIPTION:
The way total joint arthroplasty is practiced continues to evolve as CMS removed total hip arthroplasty (THA) from the inpatient-only list and added total knee arthroplasty (TKA) to the ASC Covered Surgical Procedures List (CPL) in 2020. Thus, surgeons must find subtle interventions that improve patient outcomes while minimizing the risk of adverse reactions. Current literature has not assessed the influence of preoperative hydration, using a complex carbohydrate drink, on the same-day discharge rate and causes for failure to launch. Considering variabilities in perioperative fluid management leading to postoperative nausea, vomiting, and dizziness, the investigators seek to reduce the incidence of these events by optimizing patients using a preoperative oral hydration protocol, reducing the length of stay, and improving same-day discharge rates.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for ambulatory total knee arthroplasty
* Candidates for ambulatory total hip arthroplasty
* Candidates for ambulatory revision knee arthroplasty (liner exchange only)
* Candidates for ambulatory revision hip arthroplasty (liner exchange only)
* Case scheduled before noon (12 pm)
* Patient agrees to same-day discharge and has a responsible adult to spend the night on the day of discharge

Exclusion Criteria:

* BMI less than 18.5 or greater than 37.0
* Patients with diabetes, chronic kidney disease, clotting disorders, or neurological conditions preventing control of the affected limb.
* Pregnant women
* Patients scheduled as ambulatory due to insurance mandates
* Patients with a history of active ischemia, significant valvular disease, significant arrhythmias, obstructive sleep apnea as per Hospital for Special Surgery guidelines, chronic opioid dependence (chronic daily opioid use for six or more months), and glomerular filtration rate < 60ml/min.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay in hours | From admission to discharge, up to 1 week
  Length of hospital stay in hours, assess by medical record.

SECONDARY OUTCOMES:
Same day discharge rate | Through study completion, an average of 3 months.
  Percentage of patients discharged successfully the day of surgery.
Number of physical therapy sessions attempted | From admission to discharge, up to 1 week.
  Number of physical therapy sessions attempted, assess by medical record.
Total distance walked | From admission to discharge, up to 1 week.
  Total distance walked during physical therapy attempts, assess by medical record.
Number of stairs climbed | From admission to discharge, up to 1 week.
  Number of stairs climbed during physical therapy attempts, assess by medical record.
Orthostatic hypotension episodes | During physical therapy attempts, from admission to discharge.
  Orthostatic hypotension episodes during physical therapy attempts, assess by medical record.
HOOS JR Score | The morning of surgery and at the first post-operative visit, up to 4 months post-op.
  This is a 6-item questionnaire that assesses patient-reported hip pain and function. Score ranges from 0-100, with 100 representing the best possible score.
KOOS JR Score | The morning of surgery and at the first post-operative visit, up to 4 months post-op.
  This is a 6-item questionnaire that assesses patient reported knee pain and function. Score ranges from -100, with 100 representing the best score possible.
VR-12 Score | The morning of surgery and at the first post-operative visit, up to 4 months post-op.
  The VR-12 is a 12-item self-reported questionnaire that assesses the patient physical and mental quality of life.
Urine osmolality | Measured preoperatively the morning of surgery.
  Urine osmolality taken preoperatively, assess by medical record.
Urine specific gravity | Measured preoperatively the morning of surgery.
  Urine specific gravity preoperatively, assess by medical record.
In-house costs | From admission to discharge, up to 1 week.
  In-house costs taking into account cost of complex carbohydrate drink vs previously published costs savings per night of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Rodriguez, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No